CLINICAL TRIAL: NCT06301893
Title: Prevalence and Mapping of Sickle Cell Trait and Disease in Uganda
Brief Title: Uganda Sickle Surveillance Study (US-3)
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Makerere University (Other); Ministry of Health, Uganda (Other Government); Mulago Hospital, Uganda (Other)
Responsible Party: Sponsor
Other Study IDs: US-3_Uganda (IRB#2013-4576)
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Biospecimen Retention: Samples With DNA — Perkin Elmer instrumentation is used for standardized isoelectric focusing tests using dried blood spots, followed by chemical elution of hemoglobin and electrophoresis using pre-cast gels. Newborn sickle genotype results with normal hemoglobin (HbA) and sickle hemoglobin (HbS) are typically FA, FAS, or FS although other variants including HbC may be detected. Calls will be made on each sample by trained technicians but also reviewed by supervisory personnel. Demographic information will be entered directly into a web-based electronic data capture system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is estimated that over 250,000 babies are born with sickle cell disease (SCD) annually in sub-Saharan Africa, and only 10% - 50% of them survive beyond five years of age. Data describing the magnitude of the sickle cell problem are lacking in most African countries. The available data on prevalence were mainly from older studies and small numbers of hospitalized patients. In Uganda, approximately 25,000 children are born with SCD but 70-80% die before their 5th birthday. Lehmann and Raper found 'sicklaemia' prevalence of 0.8% and 45% in the Sebei and Bambaa ethnic groups, respectively. A recent study found a SCT and SCD prevalence of 3% - 19% and 0% - 3%, respectively but this study addressed only 5 of Uganda's 111 districts and used a small convenience sample of children aged 6 - 60 months. The objective of this study is to determine the prevalence and map out the burden of SCT and SCD in Uganda.

DETAILED DESCRIPTION:
The investigators propose a cross-sectional study of sickle cell trait (SCT) and disease in all districts of Uganda using dried blood spots (DBS) collected from HIV exposed babies over a 12-month period. About 90,000 DBS samples collected from HIV exposed children from all districts of Uganda from February 2014 to March 2015 will be analyzed. Follow-up analysis will occur on up to 1,000,000 samples collected during 2015 - 2030 based on surveillance findings and secondary objectives. The study will be conducted at the Central Public Health (CPHL) in Kampala where the samples from across the country are collected for PCR testing. The investigators will perform hemoglobin analysis using isoelectric focusing (IEF). The overall prevalence and the prevalence by district of SCT and SCD will be determined. Geospatial mapping will be performed using a specialized software program to produce a map illustrating the prevalence of SCT and SCD throughout the country and allow associations between sickle cell trait/disease with either malaria prevalence or HIV co-morbidity. Further analysis of sickle cell disease or hemoglobin variants will be conducted using HPLC and DNA-based techniques.

ELIGIBILITY:
Inclusion Criteria:

* Up to 1,000,000 samples may be collected during 2015 - 2030 following primary analysis based on surveillance findings.

Exclusion Criteria:

* Repeat samples on the same individuals during the study period will be excluded.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All Dried Blood Spot (DBS) samples collected from HIV exposed infants from all districts of Uganda from approximately February 2014 to March 2015 will be included in the primary analysis. Up to 1,000,000 additional samples may be collected during 2015 - 2030 following primary analysis based on surveillance findings.
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2013-09-07 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HbSS and HbA | February 2014 to March 2015
  Incidence of sickle cell disease (HbSS) and sickle cell trait (HbA)

SECONDARY OUTCOMES:
Incidence of HbSS and HbA | March 2015 - March 2030
  Incidence of sickle cell disease (HbSS) and sickle cell trait (HbA)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Grace Ndeezi, MBChB, MMed, PhD, Principal Investigator — Department of Pediatrics & Child Health College of Health Sciences Makerere University
Locations (4):
- Uganda (4):
  - Makerere University, Kampala
  - Minister of Health, Kampala
  - National Coordinator EID Program, Kampala
  - Sickle Cell Clinic Department of Pediatrics & Child Health Mulago Hospital, Kampala